CLINICAL TRIAL: NCT03294967
Title: Effect of Caffeine on Ocular Circulation in High Myopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Andrew KC Lam, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSEARS20170613002
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: High Myopia; Choroid
Keywords: High Myopia; Caffeine; Choroidal Thickness; Choroidal Volume; Optical Coherence Tomography; Optical Coherence Tomography Angiography
MeSH Terms: interventions — Caffeine; Vitamin E

STUDY DESIGN:
Intervention Model Description: This will be a crossover study. Each subject is required to consume 200mg caffeine capsule and 200IU vitamin E control capsule, as control, in two different visits. The two visits will be randomized, with a washout period of at least one week.
Who Masked: Participant
Masking Description: Participants will not see the label of the capsule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caffeine (Active Comparator): To determine the effect of caffeine on ocular circulation in high myopes by consuming 200 mg caffeine capsule
  Interventions: Dietary Supplement: Caffeine
- Vitamin E (Placebo Comparator): To determine the effect of caffeine on ocular circulation in high myopes by consuming and 200 International Unit vitamin E control capsule, as control
  Interventions: Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Caffeine — As in group descriptions
  Arms: Caffeine
Dietary Supplement: Vitamin E — As in group descriptions
  Arms: Vitamin E

SUMMARY:
To investigate the effect of caffeine on ocular circulation by using Optical Coherence Tomography and Optical Coherence Tomography Angiography. This study will evaluate blood supply to the inner and outer retina after consumption of 200mg caffeine capsule, in particular its effect in high myopes.

DETAILED DESCRIPTION:
Caffeine could cause vasoconstriction. Previous studies revealed a reduction of retinal blood vessels diameter, a decrease in macular blood flow, and a decrease in blood velocity of optic nerve. Research devices, such as laser speckle tissue circulation analyzer and blue field simulation technique, were used in previous studies.

With an advancement of technology such as optical coherence tomography (OCT), choroidal thickness can be measured, which indicates blood supply to outer retina. In addition, superficial retinal vasculature can be measured using optical coherence tomography angiography (OCTA).

Previous studies found that subfoveal choroidal thickness declined with increase in myopia. A negative association between subfoveal choroidal thickness and axial length was also found. A recent study found a negative association between retinal vessel density with axial length in Chinese myopes using OCTA. Therefore, caffeine consumption may further make high myopes prone to ocular diseases development due to poor ocular circulation.

The current study will use OCTA to measure the superficial retinal vasculature and OCT to measure choroidal thickness and choroidal volume of high myopes after consumption of caffeine capsule.

Statistical analysis

Normality of data will be assessed. The effect of caffeine on choroidal thickness, choroidal volume, vessel density, and perfusion density of superficial retinal layers will be analysed using repeated-measures ANOVA (co-variates) to compare baseline data and that after caffeine consumption at various time points. If significant difference is obtained, post hoc tests will be conducted to compare results from various time points with the baseline data. Difference between different age groups will be compared using unpaired t-test or Mann Whitney test, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error should be at least -6 Diopters or lower (spherical equivalent)
* Best corrected visual acuity of at least 6/6
* Non-smoker

Exclusion Criteria:

- Diagnosed with any ocular diseases and systemic diseases

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Choroidal thickness | Within 4 hours
  Choroidal thickness measured by the optical coherence tomography

SECONDARY OUTCOMES:
Retinal vessel density | Within 4 hours
  Superficial retinal vessel density measured by OCTA

CONTACTS AND LOCATIONS:
Overall Officials: Kwok Cheung Andrew Lam, PhD, Principal Investigator — The Hong Kong Polytechinc University
Locations (1):
- School of optometry, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No